CLINICAL TRIAL: NCT00571623
Title: Automated Chest Physiotherap to Improve Outcomes in Neurocritical Care: An Intracranial Pressure Study
Brief Title: Automated Chest Physiotherapy to Improve Outcomes in Neuro
Acronym: ACTION-ICP
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Neuroscience Nursing Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00001842
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2008-08

CONDITIONS: Brain Injury; Intracranial Hypertension
Keywords: Brain Injury; Intracranial hypertension; Human subjects; Nursing care
MeSH Terms: conditions — Brain Injuries; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All subjects act as their own contral
  Interventions: Other: Chest Physiotherapy

INTERVENTIONS:
Other: Chest Physiotherapy — 10-minutes of chest physiotherapy using programmed parameters that are components of the specialty beds used in ICU

SUMMARY:
Following current standard-of-care, subjects data (brain pressure) will be recorded for 1 hour and include 10-minutes of data during which the subject recieves chest physiotherapy (CPT). The hypothesis is that CPT is not harmful to brain pressure.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effect of chest physiotherapy (CPT) on intracranial pressure (ICP). Because CPT is a normal part of the routine care provided to patients in the neurocritical care unit (NCU) this is an observational study of current practice.

1. The purpose of this study is to examine the effect of chest physiotherapy (CPT) on intracranial pressure (ICP). Because CPT is a normal part of the routine care provided to patients in the neurocritical care unit (NCU) this is an observational study of current practice.
2. The study will include only patients who currently have intracranial pressure monitoring devices in place (intraventricular and intraparenchymal). The study will last 1-hour and all subjects in the study will receive 10-minutes of CPT. The 10-minute CPT episode will be randomly assigned to occur 10, 20, 30 or 40-minutes into the study.
3. ANCOVA using SAS will be used to explore for within and between group differences in ICP. This study observes current standard practice, there are no additional risks to the subject.

ELIGIBILITY:
Inclusion Criteria:

* documented episode of elevated ICP ICP monitoring in situ neurological/neurosurgical diagnosis currently on a specialy bed

Exclusion Criteria:

* spinal cord injury such that CPT is not desired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 subjects with a neurological diagnosis and current ICP in situ.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Intracranial pressure | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: DaiWai M Olson, Phd RN CCRN, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Mission Hospital, Mission Viejo, California
  - Duke University, Durham, North Carolina
  - WakeMed Hospital, Raleigh, North Carolina

REFERENCES:
- [Background] Elf K, Nilsson P, Enblad P. Outcome after traumatic brain injury improved by an organized secondary insult program and standardized neurointensive care. Crit Care Med. 2002 Sep;30(9):2129-34. doi: 10.1097/00003246-200209000-00029. PMID 12352052
- [Background] Grap MJ, Munro CL. Preventing ventilator-associated pneumonia: evidence-based care. Crit Care Nurs Clin North Am. 2004 Sep;16(3):349-58, viii. doi: 10.1016/j.ccell.2004.03.005. PMID 15358383
- [Background] Olson DM, Thoyre SM, Turner DA, Bennett S, Graffagnino C. Changes in intracranial pressure associated with chest physiotherapy. Neurocrit Care. 2007;6(2):100-3. doi: 10.1007/s12028-007-0015-y. PMID 17522792
- [Background] Littlejohns L, Bader MK. Prevention of secondary brain injury: targeting technology. AACN Clin Issues. 2005 Oct-Dec;16(4):501-14. doi: 10.1097/00044067-200510000-00007. PMID 16269895
- [Background] Bader MK, Palmer S. Keeping the brain in the zone. Applying the severe head injury guidelines to practice. Crit Care Nurs Clin North Am. 2000 Dec;12(4):413-27. PMID 11855245
- [Background] Olson DM, Graffagnino C. Consciousness, coma, and caring for the brain-injured patient. AACN Clin Issues. 2005 Oct-Dec;16(4):441-55. doi: 10.1097/00044067-200510000-00003. PMID 16269891
- [Background] Arbour R. Aggressive management of intracranial dynamics. Crit Care Nurse. 1998 Jun;18(3):30-40; quiz 41-2. No abstract available. PMID 9677936